CLINICAL TRIAL: NCT00959504
Title: VeraCode Genotyping Test for Factor V and Factor II on the BeadXpress System
Brief Title: Detection of Factor V Leiden G1691A and Factor II (Prothrombin) G20210A Point Mutations in DNA
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Responsible Party: Don Ellis, Sr. Director of Quality, Illumina
Other Study IDs: ILMN001
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Detection and Genotyping of Factor V and Factor II Point Mutations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
As an external validation test of the performance of the VeraCode Genotyping Test for Factor V and Factor II on the BeadXpress System, clinical trials will be conducted at three sites. This study will assess genotyping accuracy as compared to bidirectional sequencing and genotyping reproducibility across variables such as user, day, and site.

ELIGIBILITY:
Inclusion Criteria:

* Patient samples will be leftover EDTA-anticoagulated whole blood from patients referred for Factor V and/or Factor II testing.

Exclusion Criteria:

* There are no applicable exclusion criteria for this test, since the genomic sequence will not vary by ethnicity, gender, age or disease. Inappropriately stored blood samples will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient samples will be leftover EDTA-anticoagulated whole blood from patients referred for Factor V and/or Factor II testing.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)